CLINICAL TRIAL: NCT01632540
Title: Investigation of the Real World Effectiveness of Beclomethasone Dipropionate (BDP) Nasal Aerosol in Perennial Allergic Rhinitis (PAR) Patients
Brief Title: Effectiveness of Beclomethasone Dipropionate Nasal Aerosol for Perennial Allergic Rhinitis
Acronym: BALANCE
Status: Completed | Type: Observational
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Collaborators: United BioSource, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: BDP-AR-401
Record Dates: First submitted 2012-06-28; First posted 2012-07-03 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Perennial Allergic Rhinitis (PAR)
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — Beclomethasone; alpha-ketoisovalerate dehydrogenase phosphatase; Nasal Sprays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Perennial Allergic Rhinitis patients
  Interventions: Drug: Beclomethasone Dipropionate (BDP) Nasal Aerosol

INTERVENTIONS:
Drug: Beclomethasone Dipropionate (BDP) Nasal Aerosol — BDP nasal aerosol 320 mcg/day will be administered to all patients as 2 sprays in each nostril once daily.
  Other Names: QNASL

SUMMARY:
This study will be a prospective observational study of "real world" BDP nasal aerosol users with PAR, with or without seasonal allergic rhinitis (SAR). Subjects will respond to monthly online surveys regarding rhinitis control, concomitant medical conditions, concomitant (non-AR) medications, current AR therapy, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 12 years or greater at time of enrollment
* Diagnosis of PAR for at least one year; and 2)a positive skin prick (ie, epicutaneous) or serum-specific IgE test within the past 2 years to a perennial allergen as appropriate for the location; and 3)PAR symptoms that are consistent with exposure to this allergen for at least one year
* Uncontrolled rhinitis symptoms at the time of assessment as confirmed by a score of 21 or less on the RCAT
* Newly prescribed BDP Nasal Aerosol (within the past 7 days but have not yet used)
* Willing and able to complete surveys in English on a computer with internet access
* Willing and able to provide informed consent prior to entering the study (or parent/caregiver/legal guardian if applicable)

Exclusion Criteria:

* Current acute or chronic sinusitis or chronic purulent nasal discharge
* Rhinitis medicamentosa or nasal structural abnormalities (including nasal polyps and clinically significant septal deviation) that significantly interfere with nasal airflow
* Acute upper respiratory infection within the past 14 days
* Used any pressurized metered-dose inhaler INS product (including BDP Nasal Aerosol and Ciclesonide Nasal Aerosol) within the past 90 days
* Used any experimental therapy for AR within the past 30 days
* Any condition which the investigator feels may interfere with the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female patients, at least 12 years of age, with a diagnosis of PAR for at least one year and who are newly prescribed BDP nasal aerosol.
Sampling Method: Non-Probability Sample
Enrollment: 824 (Actual)
Dates: Start 2012-07; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change in Rhinitis Control Assessment Test (RCAT) Score | Baseline and 6 months
  The RCAT will be completed each month and uses a one-week recall period. This questionnaire has six items that ask about nasal and other allergy symptoms and the control of these symptoms. Each question is responded to on a scale of 1-5. The responses are summed to evaluate a total score. A higher score (22-30) indicates that symptoms are well controlled. A lower score (5-21) indicates that rhinitis symptoms are not well controlled.

SECONDARY OUTCOMES:
Change in the Abbreviated Treatment Satisfaction Questionnaire for Medication (TSQM-9) score | Baseline and 6 months
  The TSQM-9 asks patients about their level of satisfaction or dissatisfaction with the medication they are taking in the study. The 3 subscales (effectiveness, convenience, global satisfaction) are rated separately, and there is no overall score. 7 questions have responses ranging from 1=extremely dissatisfied/difficult/inconvenient to 7=extremely satisfied/easy/convenient. 2 questions have responses ranging from 1=not at all confident/certain to 5=extremely confident/certain. Higher scores indicate greater satisfaction with the medication.
Change in the Work Productivity and Activity Impairment Questionnaire plus Classroom Impairment Questions: Allergy-specific (WPAI-CIQ-AS) score | Baseline and 6 months
  The WPAI-CIQ-AS is a 9-item, patient-reported scale that asks about the amount of time lost from work or academic classes due to allergies, as well as the impact of allergies on performing work in the workplace or in school or attending classes. It also asks about the effect of allergies on other usual daily activities. All questions ask for recall of the last 7 days. Outcomes are expressed as impairment percentages, with higher scores indicating greater impairment and less productivity.
Change in the Pittsburgh Sleep Quality Index (PSQI) score | Baseline and 6 months
  The PSQI is a self-rated questionnaire which assesses sleep quality and disturbances over a 1 month interval. 19 items generate 7 "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, daytime dysfunction. The scores of these components yield a "global score". A global score of 5 or greater indicates a poor sleeper.
Change in the Mini Rhinoconjunctivitis Quality of Life Questionnaire (MiniRQLQ) score | Baseline and 6 months
  This 14-item scale covers 5 domains: activity limitations, practical problems, nose symptoms, eye symptoms, other symptoms. Responses range from 0=not troubled to 6=extremely troubled. 5 component scores and a global score are calculated. Higher scores indicate being more troubled as a result of nose/eye symptoms during the past week.
Change in overall healthcare utilization | Baseline and 6 months
  Medical resources include in-patient care (hospitalizations, days of hospitalization), emergency room, and out-patient visits to physicians and other healthcare providers. The health services utilization survey asks for a 3 month recall and will be completed at baseline and months 3, 6, 9, and 12.
Change in number of non-intranasal corticosteroids (INS) medications for allergic rhinitis (AR) | Baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark Lepore, MD, Principal Investigator — Teva Pharmaceutical Industries, Ltd.
Locations (46):
- United States (46):
  - Teva Investigational Site 024, Little Rock, Alaska
  - Teva Investigational Site 028, Phoenix, Arizona
  - Teva Investigational Site 003, Encinitas, California
  - Teva Investigational Site 042, Fresno, California
  - Teva Investigational Site 006, Los Angeles, California
  - Teva Investigational Site 017, Orange, California
  - Teva Investigational Site 007, Palmdale, California
  - Teva Investigational Site 021, Paramount, California
  - Teva Investigational Site 040, Redwood City, California
  - Teva Investigational Site 014, Tallahassee, Florida
  - Teva Investigational Site 010, Tamarac, Florida
  - Teva Investigational Site 038, Albany, Georgia
  - Teva Investigational Site 031, Lawrenceville, Georgia
  - Teva Investigational Site 035, Savannah, Georgia
  - Teva Investigational Site 043, Fort Mitchell, Kentucky
  - Teva Investigational Site 034, Owensboro, Kentucky
  - Teva Investigational Site 033, Mandeville, Louisiana
  - Teva Investigational Site 004, Bethesda, Maryland
  - Teva Investigational Site 037, Novi, Michigan
  - Teva Investigational Site 026, Omaha, Nebraska
  - Teva Investigational Site 002, Brick, New Jersey
  - Teva Investigational Site 019, Corning, New York
  - Teva Investigational Site 018, New York, New York
  - Teva Investigational Site 039, Niagara Falls, New York
  - Teva Investigational Site 011, High Point, North Carolina
  - Teva Investigational Site 027, Winston-Salem, North Carolina
  - Teva Investigational Site 030, Winston-Salem, North Carolina
  - Teva Investigational Site 013, Toledo, Ohio
  - Teva Investigational Site 022, Ashland, Oregon
  - Teva Investigational Site 016, Eugene, Oregon
  - Teva Investigational Site 032, Havertown, Pennsylvania
  - Teva Investigational Site 025, Normal Square, Pennsylvania
  - Teva Investigational Site 012, Pittsburgh, Pennsylvania
  - Teva Investigational Site 023, Upland, Pennsylvania
  - Teva Investigational Site 015, Dallas, Texas
  - Teva Investigational Site 029, Dallas, Texas
  - Teva Investigational Site 009, Fort Worth, Texas
  - Teva Investigational Site 020, Houston, Texas
  - Teva Investigational Site 041, San Antonio, Texas
  - Teva Investigational Site 044, San Antonio, Texas
  - Teva Investigational Site 046, San Antonio, Texas
  - Teva Investigational Site 001, Waco, Texas
  - Teva Investigational Site 005, Murray, Utah
  - Teva Investigational Site 045, Newport News, Virginia
  - Teva Investigational Site 008, Puyallup, Washington
  - Teva Investigational Site 036, Greenfield, Wisconsin